CLINICAL TRIAL: NCT04188340
Title: Effect of Su-Man Formula Massage Oil Acupressure on Sleep Quality and Anxiety in Patients With Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMUH107-REC1-031
Record Dates: First submitted 2018-05-14; First posted 2019-12-05 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: Insomnia
Keywords: Su-Man formula massage oil; Acupressure; Meridian energy; Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Patients with insomnia divided into two groups, each group is 20 patients as follows: 1) control group, using sweet al mond o il apply to GV20, GV24 SP6 , HT7 and PC6 acupoints, and massage for 10 times before sleep continuously 28 days; 2) treatment group, using Su Man formula m assage oil apply to GV20, GV24 , SP6 , HT7 and PC6 acupoints, and massage for 10 times before sleep cont inu ously 28 days.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Placebo Comparator): using bergamot massage oil apply to GV20, GV24 SP6, HT7 and PC6 acupoints, and massage for 20 times before sleep continuously 28 days
  Interventions: Behavioral: Su-Man formula massage oil
- test group (Experimental): using Su-Man formula massage oil ap-ply to GV20, GV24, SP6, HT7 and PC6 acupoints, and massage for 20 times before sleep continuously 28 days
  Interventions: Behavioral: Su-Man formula massage oil

INTERVENTIONS:
Behavioral: Su-Man formula massage oil — bergamot massage oil:dilute bergamot essential oil(0.5%) with almond oil Su-Man formula massage oil: mixed 4 different essential oil include bergamot, red mandarin, petit grain bigarade, spikenard and diluted with almond oil 5%.
  Other Names: bergamot massage oil

SUMMARY:
The present study predict that Su-Man formula massage oil acupressure can improved sleep quality.

DETAILED DESCRIPTION:
About 7% person in general population became as insomnia every year, and that has 30% person due to insomnia induces other symptoms such as anxiety. In addition, the incidence of insomnia in the female is 50% more than in the male. Insomnia belong to the scope of bù-mèi in traditional Chinese Medicine (TCM). TCM consider that the cause of insomnia is due to unbalance between yin and yang, and acupressure can treat insomnia. Several studies report that aromatherapy can enhance sleepy. Therefore, the purpose of the present study was to assess the therapeutic effect of Su-Man formula massage oil associates with acupressure on sleepy quality and anxiety lysis. A total 40 patients with insomnia divided into two groups, each group is 20 patients as follows: 1) control group, using bergamot massage oil apply to GV20, GV24 SP6, HT7 and PC6 acupoints, and massage for 10 times before sleep continuously 28 days; 2) test group, using Su-Man formula massage oil ap-ply to GV20, GV24, SP6, HT7 and PC6 acupoints, and massage for 10 times before sleep continuously 28 days. The primary outcome measurement is the Chinese version of Insomnia Severity In-dex(ISI-C), Pittsburgh Sleep Quality Index (CPSQI), and Beck Anxiety Inventory(BAI); The secondary outcome measure is the changes of meridian energy.

ELIGIBILITY:
Inclusion Criteria:

* Women who has poor sleep status attaining a score of 5 on the Chinese Pittsburgh Sleep Quality Index
* 20-50 years

Exclusion Criteria:

* having asthma or any diseases involving notable organ damage (e.g., heart, lungs, liver, or kidney failure or severe olfactory dysfunction)
* being pregnant
* being breastfeeding
* have reached menopause
* taking any medicine for improving sleep or anxiolytic drugs
* be allergic to the oil that this study used.
* having skin problem over the applying area,
* having smoking and alchol drinking habit
* inability to participate in the full course of the intervention courses

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 38 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2019-04-02 (Actual); Study Completion 2019-04-02 (Actual)

PRIMARY OUTCOMES:
Chinese version of Pittsburgh Sleep Quality Index | 5mins
  Evaluate the sleep quaility of participants

SECONDARY OUTCOMES:
M.E.A.D (Meridian Energy Analysis Device) | 10mins
  The instrument mainly detects 24 representative points of the twelve meridians around the human body. The bioelectrical resistance of each meridian is measured by the test rod to evaluate the conductivity of each meridian, and the physiology of the subject is analyzed by computer. situation.
Chinese version of Insomnia Severity Index | 5mins
  Evaluate the sleep quaility
Chinese version of Beck Anxiety Inventory | 5mins
  measuring the severity of anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Liang Hsieh, PhD, Principal Investigator — China Medical University, China
Locations (1):
- ZEN chinese medicine clinic, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No